CLINICAL TRIAL: NCT03220750
Title: University Hospital Advanced Age Pregnant Cohort
Acronym: UNIHOPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Peking University Third Hospital (Other); Peking University First Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Shengjing Hospital (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); West China Second University Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); Beijing Obstetrics and Gynecology Hospital (Other); Tongji Hospital (Other); Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Jianmeng Liu, Prof., Peking University
Other Study IDs: 2016YFC1000401
Record Dates: First submitted 2017-07-12; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Advanced Maternal Age Pregnancy; High Risk Pregnancy; Perinatal Death; Maternal Death; Various Pregnancy Complications; Stillbirth and Fetal Death; Abortion, Spontaneous
MeSH Terms: conditions — Perinatal Death; Maternal Death; Stillbirth; Fetal Death; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The University Hospital Advanced Age Pregnant (UNIHOPE) Cohort is the major part of the National Key Research and Development Program on Reproductive Health & Major Birth Defects Control and Prevention Project, which is funded by the Ministry of Science and Technology of China. The Project is led by Prof. Zhao Yangyu, from the Department of Gynecology & Obstetrics, Peking University Third Hospital, and the UNIHOPE cohort is led by Prof. Jian-meng Liu, the Co-PI of the Project.

DETAILED DESCRIPTION:
The UNIHOPE Cohort is set up to provide comprehensive evidence for the prevention and treatment of gestational complications in pregnant women with advanced maternal age, and therefore, to meet the growing clinical challenges of increasing pregnant women with advanced age in the two-child era. The UNIHOPE Cohort is planning to recruit 22,000 pregnant women aged ≥35 years from 9 large obstetrical center of major University-affiliated Hospitals across China, between July 2016 and December 2020. All women will be enrolled prior to 14 wks of gestation, followed up at 24-28 wks, 32-34 wks of gestation, delivery, and 42 days postpartum. Data including demographics, medical history, reproductive history, prenatal health care, gestational complications, and pregnancy and birth outcomes will be collected via electronic data capture system. Venous blood of the pregnant women will be collected at enrollment and each follow-up visit during pregnancy, and placental tissue, cord blood and hair of the newborn will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Female aged ≥ 35 years
* Less than 14 gestational weeks
* Planning to receive prenatal healthcare and delivery service at the study hospital

Exclusion Criteria:

* Inability to provide informed consent
* Women with mental disorders

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The UNIHOPE Cohort is a prospective cohort study that will enroll ~22000 pregnant women aged 35 years and over from 9 large obstetrical center of University-Affiliated Hospitals. These hospitals locate at 7 supercities (Beijing, Shanghai, Guangdong, Shenyang, Wuhan, Chongqing and Chengdu) of China. Pregnant women who are planning to recieve prenatal healthcare and delivery in those hospitals are potential candidates for the study.
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major gestational complications and adverse pregnancy outcomes in pregnant women with the advanced age, for a singleton or twin and higher order multiple gestation | At enrollment, 24-28 weeks, 32-34 weeks of gestation, delivery, and 42 days postpartum
  Gestational diabetes mellitus, hypertensive disease of pregnancy, uterine scar pregnancy, placenta previa, preterm delivery, postpartum hemorrhage, low birth weight, spontaneous abortion, stillbirth, perinatal death

SECONDARY OUTCOMES:
Maternal death | At 24-28 weeks, 32-34 weeks of gestation, delivery, and 42 days postpartum
  Deaths during pregnancy or less than 42 days after termination of pregnancy.
The rate of cesarean delivery | At delivery
  Cesarean rate is defined as the number of cesarean delivery divided by the number of live births.
Gestational duration | At enrollment, delivery
  The number of weeks from the first day of the woman's last recorded menstrual period to the day of delivery deaths occurring within 28 days.
Birth weight | At delivery
  Every newborn's weight will be measured twice, but if the difference between the two measurement results is more than 0.1 kg, it will be measured for the third time, Low birth weight was defined as birth weight <2500 g.
Birth length | At delivery
  Every newborn's length will be measured twice, but if the difference between the two measurement results is more than 0.1 kg, it will be measured for the third time.

CONTACTS AND LOCATIONS:
Overall Officials: Yangyu Zhao, PhD, Study Chair — Peking University Third Hospital; Jian-meng Liu, PhD, Principal Investigator — Peking University
Locations (9):
- China (9):
  - Peking University First Hospital, Beijing
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - West China Second University Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Laopaiboon M, Lumbiganon P, Intarut N, Mori R, Ganchimeg T, Vogel JP, Souza JP, Gulmezoglu AM; WHO Multicountry Survey on Maternal Newborn Health Research Network. Advanced maternal age and pregnancy outcomes: a multicountry assessment. BJOG. 2014 Mar;121(Suppl 1):49-56. doi: 10.1111/1471-0528.12659. PMID 24641535
- [Background] Ngowa JD, Ngassam AN, Dohbit JS, Nzedjom C, Kasia JM. Pregnancy outcome at advanced maternal age in a group of African women in two teaching Hospitals in Yaounde, Cameroon. Pan Afr Med J. 2013 Apr 7;14:134. doi: 10.11604/pamj.2013.14.134.2315. Print 2013. PMID 23734279
- [Background] Carolan M. Maternal age >/=45 years and maternal and perinatal outcomes: a review of the evidence. Midwifery. 2013 May;29(5):479-89. doi: 10.1016/j.midw.2012.04.001. Epub 2012 Nov 16. PMID 23159159
- [Background] Khalil A, Syngelaki A, Maiz N, Zinevich Y, Nicolaides KH. Maternal age and adverse pregnancy outcome: a cohort study. Ultrasound Obstet Gynecol. 2013 Dec;42(6):634-43. doi: 10.1002/uog.12494. PMID 23630102
- [Background] Lisonkova S, Potts J, Muraca GM, Razaz N, Sabr Y, Chan WS, Kramer MS. Maternal age and severe maternal morbidity: A population-based retrospective cohort study. PLoS Med. 2017 May 30;14(5):e1002307. doi: 10.1371/journal.pmed.1002307. eCollection 2017 May. PMID 28558024
- [Background] Cleary-Goldman J, Malone FD, Vidaver J, Ball RH, Nyberg DA, Comstock CH, Saade GR, Eddleman KA, Klugman S, Dugoff L, Timor-Tritsch IE, Craigo SD, Carr SR, Wolfe HM, Bianchi DW, D'Alton M; FASTER Consortium. Impact of maternal age on obstetric outcome. Obstet Gynecol. 2005 May;105(5 Pt 1):983-90. doi: 10.1097/01.AOG.0000158118.75532.51. PMID 15863534
- [Background] Lisonkova S, Janssen PA, Sheps SB, Lee SK, Dahlgren L. The effect of maternal age on adverse birth outcomes: does parity matter? J Obstet Gynaecol Can. 2010 Jun;32(6):541-548. doi: 10.1016/S1701-2163(16)34522-4. PMID 20569534
- [Background] Niessen K, Werner-Bierwisch T, Metzing S, Sayn-Wittgenstein FZ. [Motherhood at the Age of 35 and Over: The Risk of Advanced Maternal Age as Perceived by Women - a Literature Study]. Z Geburtshilfe Neonatol. 2017 Jun;221(3):111-121. doi: 10.1055/s-0043-104864. Epub 2017 Jun 30. German. PMID 28666302
- [Background] Taghizadeh Z, Cheraghi MA, Kazemnejad A, Pooralajal J, Aghababaei S. Difference in Perception of Pregnancy Risk in Two Maternal Age Groups. J Clin Diagn Res. 2017 May;11(5):QC09-QC12. doi: 10.7860/JCDR/2017/23661.9915. Epub 2017 May 1. PMID 28658853
- [Background] Jolly M, Sebire N, Harris J, Robinson S, Regan L. The risks associated with pregnancy in women aged 35 years or older. Hum Reprod. 2000 Nov;15(11):2433-7. doi: 10.1093/humrep/15.11.2433. PMID 11056148
- [Derived] Yin S, Zhou Y, Zhao C, Yang J, Yuan P, Zhao Y, Qi H, Wei Y. Association of Paternal Age Alone and Combined with Maternal Age with Perinatal Outcomes: A Prospective Multicenter Cohort Study in China. J Epidemiol Glob Health. 2024 Mar;14(1):120-130. doi: 10.1007/s44197-023-00175-4. Epub 2024 Jan 8. PMID 38190051